CLINICAL TRIAL: NCT00949312
Title: Ultrastaging of Early Colon Cancer
Brief Title: Studying Lymph Nodes in Patients With Stage II Colon Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Saint John's Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000649763; UCLA-0809064; BILA-UECC-0107; IRB# 08-09-064-02
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Colorectal Cancer
Keywords: stage II colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Paraffin-embedded primary tumor and lymph node sections
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stage II unresected Colon Cancer
  Interventions: Genetic: RNA marker analysis of lymph node and primary tumors; Genetic: microarray profiling of primary tumors; Genetic: reverse transcriptase-polymerase chain reaction of lymph node specimens; Other: diagnostic laboratory RNA and DNA biomarker analysis of primary tumors; Procedure: regional lymph node dissection; Other: lymph node staining for H&E and pancytokeratin IHC

INTERVENTIONS:
Genetic: RNA marker analysis of lymph node and primary tumors
Genetic: microarray profiling of primary tumors
Genetic: reverse transcriptase-polymerase chain reaction of lymph node specimens
Other: diagnostic laboratory RNA and DNA biomarker analysis of primary tumors
Procedure: regional lymph node dissection
Other: lymph node staining for H&E and pancytokeratin IHC

SUMMARY:
RATIONALE: Diagnostic procedures that look for micrometastases in lymph nodes removed during surgery for colon cancer may help doctors learn the extent of disease.

PURPOSE: This phase I trial is studying lymph nodes in patients with stage II colon cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether the immunohistochemical and molecular presence of micrometastases in ≥ 12 lymph nodes removed during en-bloc resection in patients with stage II colon cancer correlates with 3-year disease-free survival.
* Evaluate the prognostic significance of molecular markers detected in the primary tumor and develop a microarray-based gene signature for stage II colon cancer.

OUTLINE: This is a multicenter study.

Tumor tissue and regional lymph node samples are collected during surgery for analysis of micrometastases and molecular markers by immunohistochemistry, qRT-PCR, MM qRT-PCR, qRDNA-PCR, and microarray profiling.

Patients are followed up periodically for 4 years after surgery.

ELIGIBILITY:
Inclusion Criteria: All of the following inclusion criteria must be met in order for the subject to be eligible.

1. Subjects must have CC detected by proctosigmoidoscopy, flexible endoscopy, or gastrograffin/barium enema, with no evidence of distant metastases within 8 weeks of enrollment.
2. Subjects with CC must have a computerized tomography (CT; at a minimum - spiral (helical) CT with 5-mm contiguous reconstruction algorithms and adequate volume (based on site-specific protocols) of oral and intravenous contrast agents) of the abdomen and pelvis and a chest x-ray or CT of the chest per standard of care, within 8 weeks prior to enrollment to rule out distant metastases. Subjects with preoperative CT scans and testing showing non-specific or non-diagnostic (equivocal) abnormalities may be eligible pending intraoperative exploration.
3. Greater than 18 years of age
4. Subjects must have a performance status ≤ 2 on the ECOG/Zubrod scale.
5. Subject is able to give informed consent, and must be willing to be followed clinically or by phone/email/mail correspondence
6. Subject must have a life expectancy of greater than 5 years not including the disease/diagnosis of CC.
7. Subject must have clinical assessment conducted by phone unless patients follow up are part of the regular clinical visits.

Exclusion Criteria: Any of the following criteria will exclude the subject from the study.

1. Subjects requiring emergent surgery (within 2 hours of presentation) to prevent a life-threatening situation or death such as those with a perforated colon, metabolically significant complete bowel obstruction or massive GI bleeding will be excluded. Subjects who do not require emergent surgery, such as those with occult bleeding or early or partial bowel obstruction will be permitted to enter.
2. Subjects with any history of Crohn's disease, chronic ulcerative colitis, or familial polyposis.
3. Discovery of distant metastases intra-operatively.
4. Subjects with history of another malignancy over the last three years (except for completely resected cervical, skin cancers or in-situ cancers - see Appendix B for a list of exempt cancers).
5. Pregnant and/or lactating women. Potentially childbearing subjects (pre-menopausal women) should undergo a pregnancy test within 7 days prior to surgery and after signing consent. Subjects found to be pregnant will be ineligible and withdrawn from the study.
6. Subjects should not be participating in another research protocol at the time of enrollment. Participation during follow-up is acceptable.
7. Systemic chemotherapy for node negative colon cancer.
8. Complete polypectomy by endoscopy
9. Less than 12 lymph nodes

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From the ambulatory cancer clinic, we will identify 300 stage II colon cancer patients eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2009-05 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (time to local or distant recurrence after resection) | 48 months
  The event to be used for DFS is time to recurrence (local or distant) after resection of colon cancer

SECONDARY OUTCOMES:
Overall survival (time to death from colorectal cancer) | 48 months
  The event to be used for DFS is time to death after resection of colon cancer

CONTACTS AND LOCATIONS:
Overall Officials: Anton J. Bilchik, MD, PhD, FACS, Principal Investigator — Saint John's Cancer Institute
Locations (2):
- United States (2):
  - John Wayne Cancer Institute, Santa Monica, California
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Protic M, Stojadinovic A, Nissan A, Wainberg Z, Steele SR, Chen DC, Avital I, Bilchik AJ. Prognostic Effect of Ultra-Staging Node-Negative Colon Cancer Without Adjuvant Chemotherapy: A Prospective National Cancer Institute-Sponsored Clinical Trial. J Am Coll Surg. 2015 Sep;221(3):643-51; quiz 783-5. doi: 10.1016/j.jamcollsurg.2015.05.007. Epub 2015 May 18. PMID 26213360